CLINICAL TRIAL: NCT04320160
Title: Structural Evaluation of Human Melanocytes After the Use of Autologous Platelet-rich Plasma (PRP) Versus Fractional Carbon Dioxide Laser (Fr:CO2 Laser) in Treatment of Vitiligo: (A Histological, Immunohistochemical and Molecular Study )
Brief Title: Evaluation of Human Melanocytes After the Use of PRP Versus Fractional CO2 Laser in Vitiligo
Acronym: PRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham ElGibaly, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 70265
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive control group (No Intervention): Include the thirty patients before any treatment
- PRP group (Active Comparator): Include fifteen patients that will recieve PRP sessions .Patients will receive six treatment sessions with one month interval for 6 months and will be followed up after 6 months.
  Interventions: Procedure: Platelet rich plasma
- Fractional CO2 group (Active Comparator): Include fifteen patients that will recieve FR: CO2 laser sessions.Patients will receive six treatment sessions with one month interval for 6 months and will be followed up after 6 months.
  Interventions: Procedure: Fractional CO2 laser

INTERVENTIONS:
Procedure: Platelet rich plasma — Eight milliliters of blood sample will be aspirated from the patient's peripheral vein, and the sample will be centrifuged at 1,500 rpm for 5 minutes.
  A 30-G needle will be used for superficial intradermal (ID) microinjections (0.1 mL per injection and space about 1 cm apart)
  Other Names: PRP
  Arms: PRP group
Procedure: Fractional CO2 laser — Fifteen lesions will be treated by Fr: CO2 laser (10,600 nm; KES Corporation, Beijing, China).
  Scanner spot size will be adjusted based on the lesion size. Density selected will be 0.6 in the static mode.
  Two passes with minimal overlap will be delivered. The laser will be applied to the vitiligo lesion and over a thin rim of healthy skin
  Other Names: Fr: CO2 laser
  Arms: Fractional CO2 group

SUMMARY:
Vitiligo is considered the most common chronic depigmentation disorder that affects around 0.5 -2% of the world population . In Africa , its prevelance is around 0.4% and 1.22 % in Assiut .

Treatment of vitiligo includes medical topical and systemic immune -suppressants ,phototherapy and surgical modalities .Despite the numerous treatment options , the treatment of choice is still controversial as the response is variable , unsatisfactory ,and requires a prolonged course. Therefore, new therapeutic approaches are required .

Platelet -rich plasma (PRP) is a treatment modality which has been used over the last several years in various medical and surgical fields . It is composed of high concentration of platelets , several growth factors and plasma proteins such as fibrin, fironectin ,vitronectin .This is hypothesized to stimulate keratinocytes and fibroblasts proliferation .

Another treatment modality is the fractional CO2 (Fr: CO2) laser .There are theories that fractional CO2 laser causes release of various types of cytokines and growth factors that can stimulate migration of melanocytes and act as mitogens for melanogenesis .

Melanogenesis is a complex process with involvement of multiple signaling pathways. Therefore, there have been extensive efforts to reveal the molecular mechanisms that control melanogenesis as the main step for treating hypopigmentary skin disorders .

There is yet very limited histopathological and molecular information about how the signaling networks are involved in the initiation , progression and also treatment of vitiligo disease.

DETAILED DESCRIPTION:
Vitiligo is considered the most common chronic depigmentation disorder that affects around 0.5 -2% of the world population .In Africa , its prevelance is around 0.4% and 1.22 % in Assiut .

Vitiligo may appear at any age and affect both sexes. It is a cosmetically disfiguring disorder characterized by formation of depigmented patches of skin and /or mucosa.It has a psychological devastating effect which could lead to low self-steam and poor body image .

Vitiligo disease has three types according to the distribution of lesions ; segmental, non-segmental and mixed vitiligo .It could be classified as progressing or stable according to the activity of the disease .

Vitiligo pathogenesis includes many theories (the combination theory). The important theories include: autoimmune destruction of melanocytes, genetic predisposition , altered redox status and free radical mediated melanocyte damage , impaired melanocyte adhesion or melanocytorrhagy and heightened sympathetic response and catecholamines/ neurotransmitter mediated melanocyte damage .

The treatment of vitiligo depends upon the clinical diagnosis and usually includes two strategies.

The first strategy aims to provide stability by arresting the progression of the active disease and therefore limiting the depigmented areas. The second strategy is repigmentation of the depigmented areas Treatment of vitiligo includes medical topical and systemic immune -suppressants ,phototherapy and surgical modalities .

First line of treatment includes topical corticosteroids ,calcineurin inhibitors and phototherapy . While the second line of treatment includes systemic corticosteroids , topical calcipotriol and excimer laser .Surgical methods include skin /single-hair grafting , autologous cultured melanocyte or epidermal suspension transplantations and immunomodulators .

Despite the numerous treatment options , the treatment of choice is still controversial as the response is variable , unsatisfactory ,and requires a prolonged course . High proportion of vitiligo patients are resistant to the treatment. Therefore, new therapeutic approaches are required .

Platelet -rich plasma (PRP) is a treatment modality which has been used over the last several years in various medical and surgical fields .It is a simple and cheap new break thorough in soft tissue healing which has attracted the attention of dermatologists in the skin rejuvenation field .

PRP is composed of high concentration of platelets (seven times the normal blood level ), several growth factors and plasma proteins such as fibrin, fironectin ,vitronectin . Growth factors are known to regulate many processes such as cell migration , proliferation and differentiation .This is hypothesized to stimulate keratinocytes and fibroblasts proliferation .

Another treatment modality is the fractional CO2 (Fr: CO2) laser which represents a new modality for skin rejuvenation based on the theory of fractional photothermolysis . It has been used in treating facial photo-aging and scars . There are theories that fractional CO2 laser causes release of various types of cytokines and growth factors that can stimulate migration of melanocytes and act as mitogens for melanogenesis .

Melanogenesis is a complex process with involvement of multiple signaling pathways. Therefore, there have been extensive efforts to reveal the molecular mechanisms that control melanogenesis as the main step for treating hyperpigmentary skin disorders .

Molecular signaling pathways include p38 Mitogen-activated protein kinase (MAPK) , c-Jun N-terminal kinase /stress -activated protein kinase (JNK/SAPK) and extracellular signal-regulated kinase (ERK). These pathways are important in regulating cell proliferation ,differentiation and apoptosis of melanocytes .

Another important signaling pathway is protein kinase B ( Akt )which is involved in the differentiation of the keratinocytes. Activation of the Akt pathway triggers the differentiation process and is sustained until reaching the last stage of keratinocytes differentiation.

There is yet very limited histopathological and molecular information about how these signaling networks are involved in the initiation , progression and also treatment of vitiligo disease.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20-60 years old
* Avoid using any other treatment modalities for vitiligo during the course of the study

Exclusion Criteria:

* Pregnant and lactating women
* local medications or laser therapy one month prior to the study
* bleeding disorders
* history of keloid formation
* photosensitivity
* seizure disorders

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2022-10-24 (Estimated)

PRIMARY OUTCOMES:
melanocyte cell quantification by light microscope | 1 year
  Punch biopsy specimens will be stained by special immunohistochemical stain of Melan A antibody marker then counting melanocyte cells per field in five non overlapping fields using NIKON camera attached to a light microscope

SECONDARY OUTCOMES:
Mean improvement score by physician (MISP) | 1 year
  MISP will be calculated by comparing the photographs. Physicians' clinical assessments will be done by two blinded dermatologists using a quartile grading scale (grade 1: <25%, no or minimal improvement; grade 2: 25%-49%, moderate; grade 3: 50%-74%, marked; grade 4: >75%-99%, excellent; and grade 5: 100%, complete)

CONTACTS AND LOCATIONS:
Overall Officials: Amal T. ELghait, Professor, Principal Investigator — Assiut University

REFERENCES:
- [Background] Kadry M, Tawfik A, Abdallah N, Badawi A, Shokeir H. Platelet-rich plasma versus combined fractional carbon dioxide laser with platelet-rich plasma in the treatment of vitiligo: a comparative study. Clin Cosmet Investig Dermatol. 2018 Nov 8;11:551-559. doi: 10.2147/CCID.S178817. eCollection 2018. PMID 30510437
- [Background] Abdel-Hafez K, Abdel-Aty MA, Hofny ER. Prevalence of skin diseases in rural areas of Assiut Governorate, Upper Egypt. Int J Dermatol. 2003 Nov;42(11):887-92. doi: 10.1046/j.1365-4362.2003.01936.x. PMID 14636205
- [Background] Kim HJ, Hong ES, Cho SH, Lee JD, Kim HS. Fractional Carbon Dioxide Laser as an "Add-on" Treatment for Vitiligo: A Meta-analysis with Systematic Review. Acta Derm Venereol. 2018 Feb 7;98(2):180-184. doi: 10.2340/00015555-2836. PMID 29110015
- [Background] Abuaf OK, Yildiz H, Baloglu H, Bilgili ME, Simsek HA, Dogan B. Histologic Evidence of New Collagen Formulation Using Platelet Rich Plasma in Skin Rejuvenation: A Prospective Controlled Clinical Study. Ann Dermatol. 2016 Dec;28(6):718-724. doi: 10.5021/ad.2016.28.6.718. Epub 2016 Nov 23. PMID 27904271
- [Background] Calautti E, Li J, Saoncella S, Brissette JL, Goetinck PF. Phosphoinositide 3-kinase signaling to Akt promotes keratinocyte differentiation versus death. J Biol Chem. 2005 Sep 23;280(38):32856-65. doi: 10.1074/jbc.M506119200. Epub 2005 Jul 21. PMID 16036919
- [Background] Bishnoi A, Parsad D. Clinical and Molecular Aspects of Vitiligo Treatments. Int J Mol Sci. 2018 May 18;19(5):1509. doi: 10.3390/ijms19051509. PMID 29783663
- [Background] Kumar R, Parsad D, Kanwar AJ, Kaul D. Altered levels of Ets-1 transcription factor and matrix metalloproteinases in melanocytes from patients with vitiligo. Br J Dermatol. 2011 Aug;165(2):285-91. doi: 10.1111/j.1365-2133.2011.10324.x. PMID 21428970
- [Background] Li L, Wu Y, Li L, Sun Y, Qiu L, Gao XH, Chen HD. Triple combination treatment with fractional CO2 laser plus topical betamethasone solution and narrowband ultraviolet B for refractory vitiligo: a prospective, randomized half-body, comparative study. Dermatol Ther. 2015 May-Jun;28(3):131-4. doi: 10.1111/dth.12202. Epub 2015 Mar 5. PMID 25753514
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Background] Picardo M, Dell'Anna ML, Ezzedine K, Hamzavi I, Harris JE, Parsad D, Taieb A. Vitiligo. Nat Rev Dis Primers. 2015 Jun 4;1:15011. doi: 10.1038/nrdp.2015.11. PMID 27189851
- [Background] Rodrigues M, Ezzedine K, Hamzavi I, Pandya AG, Harris JE; Vitiligo Working Group. Current and emerging treatments for vitiligo. J Am Acad Dermatol. 2017 Jul;77(1):17-29. doi: 10.1016/j.jaad.2016.11.010. PMID 28619557
- [Background] Wrotniak M, Bielecki T, Gazdzik TS. Current opinion about using the platelet-rich gel in orthopaedics and trauma surgery. Ortop Traumatol Rehabil. 2007 May-Jun;9(3):227-38. English, Polish. PMID 17721419
- [Background] Zhang Y, Cai Y, Shi M, Jiang S, Cui S, Wu Y, Gao XH, Chen HD. The Prevalence of Vitiligo: A Meta-Analysis. PLoS One. 2016 Sep 27;11(9):e0163806. doi: 10.1371/journal.pone.0163806. eCollection 2016. PMID 27673680